CLINICAL TRIAL: NCT01940120
Title: A Study of the Evalve® Cardiovascular Valve Repair (MitraClip®) System Endovascular Valve Edge-to-Edge REpair STudy (EVEREST II) EVEREST II High Risk Registry
Brief Title: EVEREST II Pivotal Study High Risk Registry (HRR)
Acronym: HRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0401A
Record Dates: First submitted 2013-09-03; First posted 2013-09-12 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency
Keywords: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency; Mitral Valve; MR; Mitral Valve Prolapse; Edge to Edge (E2E); Alfieri Technique; MitraClip; Functional MR; Degenerative MR; Echocardiogram; Coronary Artery Disease (CAD); Heart Failure; Heart Attack; EVEREST; EVEREST I; EVEREST II; REALISM
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Coronary Artery Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Risk Registry Arm (Experimental): Includes patients with a predicted procedural mortality of 12% or higher. The high risk registry arm of the study is powered to show superiority of safety of treatment with the MitraClip compared to mitral valve surgery. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip implant.
  Interventions: Device: Percutaneous mitral valve repair using MitraClip implant

INTERVENTIONS:
Device: Percutaneous mitral valve repair using MitraClip implant — Procedure/Surgery: Mitral valve repair or replacement surgery Repair or replacement of mitral valve
  Other Names: MitraClip; MitraClip Implant

SUMMARY:
Prospective, multi-center, single arm registry. Clinical follow-up at discharge, 30 days, 6, 12, 18 and 24, months, and 3, 4 and 5 years.

Concurrent Control (CC) group identified retrospectively from the patients screened for the HRR who did not enroll; patient survival determined at 12 months. NCT00209274 (EVEREST II RCT) Intended use Percutaneous reduction of clinically significant mitral regurgitation in symptomatic patients who are considered to be high risk for operative mortality (high surgical risk).

DETAILED DESCRIPTION:
The EVEREST II HRR is a single-arm prospective, multicenter clinical trial enrolling high surgical risk patients of the EVEREST II study (NCT00209274).

Patients were considered high surgical risk if either their Society of Thoracic Surgery (STS) predicted operative mortality risk was ≥ 12%, or the surgeon investigator determined the patient to be high risk (≥ 12% predicted operative mortality risk) due to the presence of, at a minimum, one of the following pre-specified risk factors:

* Porcelain aorta or mobile ascending aortic atheroma
* Post-radiation mediastinum
* Previous mediastinitis
* Functional MR with ejection fraction (EF) < 40%
* Over 75 years old with EF < 40%
* Prior re-operation with patent grafts
* Two or more prior chest surgeries
* Hepatic cirrhosis
* Three or more of the following STS high risk factors:

  i. Creatinine > 2.5 mg/dL ii. Prior chest surgery iii. Age over 75 iv. EF < 35%

Upon completion of enrollment in the HRR, a process was initiated to ensure patient consent to participate in a Concurrent Control (CC) group was in place. Patients were identified to determine survival through 12 months with current standard of care treatment.CC patients were derived from a cohort of patients screened for enrollment in the HRR,yet did not enroll. All patients had moderate-to-severe (3+) or severe (4+) MR based on transthoracic echocardiography (TTE). To be considered eligible for inclusion in the CC group, the patient had to be classified as high surgical risk using the same criteria used for the HRR. Upon follow-up with the clinical sites, it was determined that some of the initially identified patients with moderate-to-severe (3+) or severe (4+) MR met the criteria for high surgical risk. Of these patients, some were not included due to; lack of Institutional Review Board (IRB) approval at the site, lack of informed consent and unable to be contacted. The remaining patients make up the CC group.

ELIGIBILITY:
Inclusion Criteria:

Candidates for the high risk arm of the study must meet all of the following inclusion criteria:

* Predicted procedural mortality risk calculated using the STS surgical risk calculator of ≥ 12% or in the judgment of the surgeon investigator the patient is considered a high risk surgical candidate due to the presence of one of the following indications:

  1. Porcelain aorta or mobile ascending aortic atheroma
  2. Post-radiation mediastinum
  3. Previous mediastinitis
  4. Functional MR with EF<40
  5. Over 75 years old with EF<40
  6. Re-operation with patent grafts
  7. Two or more prior chest surgeries
  8. Hepatic cirrhosis i Three or more of the following STS high risk factors: i) Creatinine > 2.5 mg/dL ii) Prior chest surgery iii) Age over 75 iv) EF<35
* Age 18 years or older.
* Symptomatic moderate to severe (3+) or severe (4+) chronic mitral regurgitation (MR) and in the judgment of the investigator intervention to reduce MR is likely to provide symptomatic relief for the patient. MR is determined as defined in Appendix A of the EVEREST II study protocol. American Society of Anesthesiologists (ASA) physical status classification of ASA IV or lower.
* The primary regurgitant jet originates from malcoaptation of the A2 and P2 scallops of the mitral valve.
* Male or Female. Female subjects of childbearing potential must have a negative pregnancy test within seven (7) days before the procedure.
* The subject or the subject's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board of the respective clinical site.
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
* Transseptal catheterization is determined to be feasible by the treating physician.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

* Evidence of an acute myocardial infarction in the prior 2 weeks of the intended treatment (defined as: Q wave or non-Q wave infarction having creatine kinase (CK) enzymes ≥ two times (2X) the upper laboratory normal limit with the presence of a Creatine Kinase MB Isoenzyme (CKMB) elevated above the institution's upper limit of normal).
* In the judgment of the Investigator, the femoral vein cannot accommodate a 24 F catheter or presence of ipsilateral deep vein thrombosis (DVT).
* Ejection fraction < 20%, and/or end-systolic dimension > 60 mm as defined in Appendix A of the EVEREST II protocol.
* Mitral valve orifice area < 4.0 cm2 as defined in Appendix A of the EVEREST II protocol.
* If leaflet flail is present:

  1. Flail Width: the width of the flail segment is greater than or equal to 15 mm, as defined in Section 4.3 and Appendix A, or
  2. Flail Gap: the flail gap is greater than or equal to 10 mm, as defined in Section 4.3 and Appendix A.
* If leaflet tethering is present:

  a). Coaptation Length: the vertical coaptation length is less than 2 mm, as defined in Section 4.3 and Appendix A.
* Leaflet anatomy which may preclude clip implantation, proper clip positioning on the leaflets or sufficient reduction in MR. This may include:
* Evidence of calcification in the grasping area of the A2 and/or P2 scallops
* Presence of a significant cleft of A2 or P2 scallops
* More than one anatomic criteria dimensionally near the exclusion limits
* Bileaflet flail or severe bileaflet prolapse
* Lack of both primary and secondary chordal support
* Hemodynamic instability defined as systolic pressure < 90 mmHg without after load reduction or cardiogenic shock or the need for inotropic support or intra-aortic balloon pump.
* Need for emergent or urgent surgery for any reason.
* Prior mitral valve leaflet surgery or any currently implanted mechanical prosthetic mitral valve.
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic diseased (i.e. noncompliant, perforated).
* History of bleeding diathesis or coagulopathy or subject will refuse blood transfusions.
* Active infections requiring current antibiotic therapy (if temporary illness, patients may enroll 2 weeks after discontinuation of antibiotics). Patients must be free from infection prior to treatment. Any required dental work should be completed a minimum of 3 weeks prior to treatment.
* Intravenous drug abuse or suspected inability to adhere to follow-up.
* Patients in whom transesophageal echocardiography (TEE) is contraindicated.
* A known hypersensitivity or contraindication to study or
* In the judgment of the Investigator, patients in whom the presence of a permanent pacemaker or pacing leads would interfere with placement of the test device or the placement of the test device would disrupt the leads.
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. [Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Feldman, M.D., Principal Investigator — Endeavor Health; Donald G Glower Jr.,, M.D., Principal Investigator — Duke University Medical Center, Department of Surgery
Locations (2):
- United States (2):
  - Evanston Northwestern Healthcare 2650 Ridge Ave., Walgreen Bldg, 3rd Floor, Cardiology, Evanston, Illinois
  - The Care Group Heart Center 10590 N. Meridian, Ste. 300, Indianapolis, Indiana

REFERENCES:
- [Derived] Ailawadi G, Lim DS, Mack MJ, Trento A, Kar S, Grayburn PA, Glower DD, Wang A, Foster E, Qasim A, Weissman NJ, Ellis J, Crosson L, Fan F, Kron IL, Pearson PJ, Feldman T; EVEREST II Investigators. One-Year Outcomes After MitraClip for Functional Mitral Regurgitation. Circulation. 2019 Jan 2;139(1):37-47. doi: 10.1161/CIRCULATIONAHA.117.031733. PMID 30586701
- [Derived] Kar S, Feldman T, Qasim A, Trento A, Kapadia S, Pedersen W, Lim DS, Kipperman R, Smalling RW, Bajwa T, Hermann HC, Hermiller JB, Lasala JM, Reisman M, Glower D, Mauri L, Whitlow P; EVEREST II Investigators. Five-year outcomes of transcatheter reduction of significant mitral regurgitation in high-surgical-risk patients. Heart. 2019 Nov;105(21):1622-1628. doi: 10.1136/heartjnl-2017-312605. Epub 2018 Aug 4. PMID 30077993
- [Derived] Wang A, Sangli C, Lim S, Ailawadi G, Kar S, Herrmann HC, Grayburn P, Foster E, Weissman NJ, Glower D, Feldman T. Evaluation of renal function before and after percutaneous mitral valve repair. Circ Cardiovasc Interv. 2015 Jan;8(1):e001349. doi: 10.1161/CIRCINTERVENTIONS.113.001349. PMID 25593120
- See also: Sponsor information — https://www.vascular.abbott/us/homepage.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who met eligibility criteria for the study and had a MitraClip procedure, whether a Device was implanted or not, were considered enrolled in the Registry. A total of 78 patients were enrolled at 35 North American sites. Screening period: Jan, 2007-2008. Enrollment period: Feb 14, 2007- Jan 30, 2008.
Period: Overall Study
Arm/Group | High Risk Registry Arm
Started | 78
Completed | 30
Not Completed | 48
Not completed — Death | 40
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (9.8)
Age, Customized [Number; unit: participants]
  18-75 years | 30
  >75 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 77
  Canada | 1
Predicted Surgical Mortality [Mean (Standard Deviation); unit: Probability percentage] — The Society of Thoracic Surgeons' risk models predict the risk of operative mortality & morbidity after adult cardiac surgery.
  Risk models were developed for nine specific endpoints, including operative mortality.Operative mortality includes both (1) all deaths occurring during the hospitalization, even if after 30 days (2) deaths occurring after discharge, but within 30 days of the procedure.
  Therefore, a patient's mortality risk score is defined as the patient's predicted risk of operative mortality as calculated by the specific operative mortality statistical model.
  Probability percentage | 18.2 (8.0)
LV Measurement [Mean (Standard Deviation); unit: mL]
  Left Ventricular End Diastolic Volume (LVEDV) | 166.5 (50.7)
  Left Ventricular End Systolic Volume (LVESV) | 79.9 (42.7)
LV Measurement [Mean (Standard Deviation); unit: cm]
  Left Ventricular Internal Diameter Diastole(LVIDd) | 5.6 (0.7)
  Left Ventricular Internal Diameter Systole (LVIDs) | 3.9 (1.1)
36-Item Short Form Health Survey (SF-36) Quality of Life [Mean (Standard Deviation); unit: scores on a scale] — The SF-36 is a multidimensional, patient-reported survey containing 36 questions on a 0-100 scale measuring physical (Physical Component Score PCS) & mental health status (Mental Component Score MCS) in relation to 8 health concepts: physical functioning, role limitations due to physical or emotional health, bodily pain, general health perceptions, vitality, social functioning, & general mental health. Higher scores represent better self-perceived health. The PCS & MCS norms for 65-75 year olds are 44 and 52, while the norms for CHF population are 31 and 46, respectively.
  scores on a scale
    Physical Health (PCS) | 31.6 (9.1)
    Mental Health (MCS) | 44.2 (12.6)
NYHA Functional Class [Number; unit: participants] — Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest & discomfort is increased with physical activity.
  participants
    NYHA Functional Class I | 0
    NYHA Functional Class II | 8
    NYHA Functional Class III | 47
    NYHA Functional Class IV | 23
Number of patients hospitalized for CHF during 12 months before enrollment [Number; unit: participants]
  Number of patients hospitalized for CHF | 33
  Number of patients not hospitalized for CHF | 45
Number of CHF events leading to hospitalizations during 12 months before enrollment [Number; unit: events] | 51
Number of hospitalization days for CHF at 12 months before enrollment [Mean (Standard Deviation); unit: days] | 6.0 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Composite Functional and Structural Measures - Freedom From Death
Description: Defined as all causes of death for the primary safety Major Adverse Event (MAE) Endpoint. Death is further divided into 2 categories:
  A. Cardiac death is defined as death due to any of the following:
  1. Acute myocardial infarction.
  2. Cardiac perforation/pericardial tamponade.
  3. Arrhythmia or conduction abnormality.
  4. Stroke within 30 days of the procedure or stroke suspected of being related to the procedure.
  5. Death due to any complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.
  6. Any death for which a cardiac cause cannot be excluded.
  B. Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 59

2. Primary Outcome: Percentage of Participants With Freedom From Death and Mitral Regurgitation (MR) >2+
Description: Kaplan-Meier estimated percentage of patients who are alive and have a mitral regurgitation severity grade of 2+ or less
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
percentage of participants
  Primary Analysis | 56.4
  Worst case Analysis | 53.8

3. Primary Outcome: Number of Participants With Clinical Measures of Benefit-New York Heart Association (NYHA) Class
Description: The major effectiveness endpoint is an assessment of multiple functional and structural measures of benefit including New York Heart Association (NYHA) Class.
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 30 days
Population: 71 out of 78 patients (at baseline) were analyzed at 30 days. There were 6 deaths prior to 30 days. So, NYHA at 30 days is missing due to death in 6 patients, and missing due to other reasons in 1 patient.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 71
Participants
  NYHA Functional Class I | 14
  NYHA Functional Class II | 38
  NYHA Functional Class III | 16
  NYHA Functional Class IV | 3

4. Primary Outcome: Number of Participants With New York Heart Association (NYHA) Class
Description: Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 12 months
Population: Of 78 total population, 54 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and 2 patients without NYHA Class assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
Participants
  NYHA Functional Class I | 18
  NYHA Functional Class II | 22
  NYHA Functional Class III | 13
  NYHA Functional Class IV | 1

5. Primary Outcome: Clinical Measures of Benefit-Quality of Life (QOL) as Measured by Short Form (SF) 36
Description: Standardized quality of life surveys allow physicians to evaluate the effectiveness of different treatment methods and the physical and psychological benefits a patient is likely to receive from a particular treatment.In the EVEREST II HRR,the patients were asked to complete the SF-36 QOL survey at baseline, 30 days and 12 months. The physical & mental function were assessed by the Physical Component Summary (PCS) score & Mental Component Summary (MCS) score. The PCS & MCS norms for 65-75 year olds are 44 and 52 respectively; and 31 & 46 for congestive heart failure (CHF) patients respectively. Each scale from the SF-36 is an algebraic sum of responses for all items in that scale.For ease of analysis each scale is then transformed to a 0-100 scale using a formula that converts the lowest & highest possible scores to 0 & 100 respectively.The scoring of the SF-36 indicates that 0% in a domain represents the poorest possible QoL & 100% indicates full QoL.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 47
score on a scale
  PCS | 36.1 (10.8)
  MCS | 48.7 (11.9)

6. Primary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: Left Ventricular End Diastolic Volume (LVEDV) as determined by the core echocardiography laboratory from a transthoracic echocardiogram (TTE).
Time Frame: 12 months
Population: Of 78 total population, 54 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and LVEDV was not done or un-evaluable in 2 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
ml | 139.7 (42.6)

7. Primary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular End Systolic Volume (LVESV) as determined by the core echocardiography laboratory from a transthoracic echocardiogram (TTE).
Time Frame: 12 months
Population: Of 78 total population, 54 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and LVESV was not done or un-evaluable in 2 patients.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
ml | 72.2 (35.8)

8. Primary Outcome: Left Ventricular (LV) Function - Internal Dimension
Description: Left Ventricular Internal Dimension in diastole (LVIDd) and Left Ventricular Internal Dimension in systole (LVIDs) as determined by the core echocardiography laboratory from a transthoracic echocardiogram (TTE).
Time Frame: 12 months
Population: Of 78 total population, 54 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and LIVDs/LVIDs evaluation was not done or un-evaluable in 2 patients.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
cm
  LV Internal Dimension diastole (LVIDd) | 5.3 (0.7)
  LV Internal Dimension systole (LVIDs) | 3.8 (1.0)

9. Primary Outcome: Number of Patients With CHF Having Hospitalization During Discharge Through 12 Months
Description: Number of patients with incidence of re-hospitalizations for CHF in the 12-months after the MitraClip implant procedure.
Time Frame: 12 months
Population: Three patients died before discharge and thus do not provide data on post-discharge hospitalizations.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
Participants | 12

10. Primary Outcome: Number of CHF Events Leading to Hospitalizations During Discharge Through 12 Months
Description: Incidence of re-hospitalizations for CHF in the 12-months after the MitraClip implant procedure.
Time Frame: 12 months
Population: Three patients died before discharge and thus do not provide data on post-discharge hospitalizations.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
Participants | 22

11. Primary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 6
Time Frame: Discharge or 30 days
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
ml | 147.9 (48.8)

12. Primary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 7
Time Frame: Discharge or 30 days
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
ml | 74.3 (40.4)

13. Primary Outcome: Left Ventricular (LV) Function - Internal Dimension
Description: as for outcome 8
Time Frame: Discharge or 30 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 76
cm
  LV Internal Dimension diastole (LVIDd) | 5.4 (0.8)
  LV Internal Dimension systole (LVIDs) | 3.9 (1.0)

14. Secondary Outcome: Number of Participants Experiencing Major Adverse Events (MAE)
Description: Combined clinical endpoint of death, myocardial infarction, reoperation for failed surgical repair or replacement, nonelective cardiovascular surgery for adverse events, stroke, renal failure, deep wound infection, ventilation for greater than 48 hours, GI complication requiring surgery, new onset of permanent atrial fibrillation, septicemia, and transfusion of 2 or more units of blood.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 21

15. Secondary Outcome: Number of Participants Experiencing Major Adverse Events
Description: as for outcome 14
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 33

16. Secondary Outcome: Procedural Freedom From In-hospital MAE
Description: Percutaneous Clip procedure or surgery with no occurrence of in-hospital MAE.
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
participants | 61

17. Secondary Outcome: Number of Participants Over 75 Years of Age With MAE
Description: as for outcome 14
Time Frame: 30 days
Population: Analysis population includes 48 patients who were aged 75 years or older in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 48
Participants | 14

18. Secondary Outcome: Number of Participants Over 75 Years of Age With MAE
Description: as for outcome 14
Time Frame: 12 months
Population: Analysis population includes 48 patients who were aged 75 years or older in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 48
Participants | 23

19. Secondary Outcome: Number of Participants Experiencing Major Vascular Complications
Description: Defined as the occurrence of any of the following resulting from the index procedure:
  * Hematoma at access site >6 cm;
  * Retroperitoneal hematoma;
  * Arterial-venous fistula;
  * Symptomatic peripheral ischemia/ nerve injury with clinical signs or symptoms lasting >24 hours;
  * Vascular surgical repair at catheter access sites;
  * Pulmonary embolism;
  * Ipsilateral deep vein thrombus; or
  * Access site-related infection requiring intravenous antibiotics and/or extended hospitalization.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

20. Secondary Outcome: Number of Participants Experiencing Major Vascular Complications
Description: as for outcome 19
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 3

21. Secondary Outcome: Number of Participants With Major Bleeding Complications
Description: Defined as procedure related bleeding that requires a transfusion of ≥2 units of blood and/or surgical intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 13

22. Secondary Outcome: Number of Participants With Major Bleeding Complications
Description: Defined as procedure related bleeding that requires a transfusion of ≥2 units of blood and/or surgical intervention.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 15

23. Secondary Outcome: Number of Participants With Non-cerebral Thromboembolism
Description: Defined as any mural thrombus or thromboembolism in the vasculature (excluding central nervous system events) confirmed by standard clinical and laboratory testing and which requires intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

24. Secondary Outcome: Number of Participants With Non-cerebral Thromboembolism
Description: as for outcome 23
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 1

25. Secondary Outcome: Number of Participants With Thrombosis
Description: Evidence of formation of an independently moving thrombus on any part of the Clip or any commercially available implant used during surgery by echocardiography or fluoroscopy. If Clip is explanted or an autopsy is performed this diagnosis should be confirmed.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

26. Secondary Outcome: Number of Participants With Thrombosis
Description: as for outcome 25
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

27. Secondary Outcome: Number of Participants With Hemolysis
Description: Defined as new onset of anemia associated with laboratory evidence of red cell destruction. Diagnosed when plasma free hemoglobin is greater than 40 mg/dL on two measures within 24 hours or on one measure if intervention is initiated based on other clinical symptoms
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

28. Secondary Outcome: Number of Participants With Hemolysis
Description: as for outcome 27
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

29. Secondary Outcome: Number of Participants With Dysrhythmias
Description: Includes all new onset atrial fibrillation and heart block requiring placement of a permanent pacemaker.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 5

30. Secondary Outcome: Number of Participants With Dysrhythmias
Description: Includes all new onset atrial fibrillation and heart block requiring placement of a permanent pacemaker.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 8

31. Secondary Outcome: Number of Participants With Endocarditis
Description: Using Duke Criteria, endocarditis can be confirmed by:
  Pathological criteria: Endocarditis is confirmed if microorganisms are identified by culture or histology in a vegetation, embolized vegetation, or an intracardiac abscess; or if pathological lesions are observed & histologically confirmed showing active endocarditis.
  Clinical criteria: Endocarditis is confirmed by the presence of 2 major criteria, 1 major plus 3 minor criteria, or 5 minor criteria. Major criteria include persistently +ve blood cultures with the presence of typical organisms for endocarditis; persistent bacteremia; evidence of endocardial involvement with positive echocardiogram with signs of oscillating vegetation, abscesses, valve perforation, new partial dehiscence of prosthetic valve or new valvular regurgitation. Minor criteria include predisposing heart condition, fever, vascular phenomena, immunologic phenomena, & positive blood culture or echocardiogram not meeting major criteria.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 0

32. Secondary Outcome: Number of Participants With Endocarditis
Description: as for outcome 31
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 1

33. Secondary Outcome: Number of Participants With Atrial Septal Defect (ASD)
Description: Occurrence of clinically significant ASD as a result of the procedure requiring intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- High Risk Registry Arm: Includes patients with a predicted procedural mortality of 12% or higher. The high risk registry arm of the study is powered to show superiority of safety of treatment with the MitraClip compared to mitral valve surgery. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip implant.
  .
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

34. Secondary Outcome: Number of Participants With Atrial Septal Defect (ASD)
Description: Occurrence of clinically significant ASD as a result of the procedure requiring intervention.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

35. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Mitral stenosis associated with a total mitral valve orifice area less than 1.5 cm2.
Time Frame: 30 days
Population: Of total 78 participants, only 72 participants were analyzed as 6 deaths within 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 72
Participants | 0

36. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Mitral stenosis associated with a total mitral valve orifice area less than 1.5 cm2.
Time Frame: 12 months
Population: Of total 78 participants, only 72 participants were analyzed because 3 patients were not implanted with a device and 3 patients died prior to discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 72
Participants | 0

37. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Mitral stenosis associated with a total mitral valve orifice area less than 1.5 cm2.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

38. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Mitral stenosis associated with a total mitral valve orifice area less than 1.5 cm2.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

39. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Mitral stenosis associated with a total mitral valve orifice area less than 1.5 cm2.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

40. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 30 days
Population: Of 78 total population, 50 participants were included in analysis population because of 6 deaths and Mitral Valve Area by planimetry was not done in 22 patients.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 50
cm^2 | 3.3 (0.9)

41. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 12 months
Population: Of 78 total population, 45 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 11 patients Mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 45
cm^2 | 3.0 (1.0)

42. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 24 months
Population: Of 78 total population, 19 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 25 patients Mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 19
cm^2 | 3.3 (0.6)

43. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 36 months
Population: Of 78 total population, 25 participants were included in analysis population because of 31 deaths within 3 years, 7 withdrawals, 1 missed visit and in 14 patients mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 25
cm^2 | 2.9 (0.8)

44. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 48 months
Population: Of 78 total population, 18 participants were included in analysis population because of 33 deaths within 4 years, 8 withdrawals, 3 missed visit and in 16 patients Mitral Valve Area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 18
cm^2 | 3.0 (0.7)

45. Secondary Outcome: Mitral Valve Area: By Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 19
cm^2 | 2.9 (0.8)

46. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 30 days
Population: Of 78 total population, 66 participants were included in analysis population because of 6 deaths and in 6 patients Mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 66
cm^2 | 2.9 (1.2)

47. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 12 months
Population: Of 78 total population, 53 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 3 patients Mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
cm^2 | 3.0 (1.2)

48. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 24 months
Population: Of 78 total population, 40 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 4 patients Mitral valve area evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 40
cm^2 | 2.8 (0.8)

49. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 35
cm^2 | 2.9 (0.8)

50. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
cm^2 | 2.8 (0.9)

51. Secondary Outcome: Mitral Valve Area: By Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
cm^2 | 2.8 (0.7)

52. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: Mitral valve area as measured by core lab echocardiography by planimetry and indexed to body surface area [MVA Index = MVA (cm^2)/BSA (m^2)].
Time Frame: 30 days
Population: Of 78 total population, 50 participants were included in analysis population because of 6 deaths and Mitral Valve Area Index by planimetry was not done in 22 patients.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 50
cm^2/m^2 | 1.7 (0.5)

53. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: as for outcome 52
Time Frame: 12 months
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 45
cm^2/m^2 | 1.6 (0.5)

54. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: as for outcome 52
Time Frame: 24 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 19
cm^2/m^2 | 1.7 (0.3)

55. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: as for outcome 52
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 25
cm^2/m^2 | 1.5 (0.4)

56. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: as for outcome 52
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 18
cm^2/m^2 | 1.5 (0.4)

57. Secondary Outcome: Mitral Valve Area Index : By Planimetry
Description: as for outcome 52
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 19
cm^2/m^2 | 1.5 (0.4)

58. Secondary Outcome: Mitral Valve Area (MVA) Index: by Pressure-Half Time Formula
Description: Mitral valve area as measured by core lab echocardiography using the pressure half-time formula and indexed to Body surface area (BSA).
  [MVA Index = MVA (cm^2)/BSA (m^2)]
Time Frame: 30 days
Population: Of 78 total population, 65 participants were included in analysis population because of 6 deaths and Mitral Valve Area Index by pressure half-time was not done in 7 patients.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 65
cm^2/m^2 | 1.6 (0.7)

59. Secondary Outcome: Mitral Valve Area Index : By Pressure Half-time Formula
Description: Mitral valve area as measured by core lab echocardiography using the pressure half-time formula and indexed to body surface area [MVA Index = MVA (cm^2)/BSA (m^2)].
Time Frame: 12 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
cm^2/m^2 | 1.6 (0.7)

60. Secondary Outcome: Mitral Valve Area Index : By Pressure Half-time Formula
Description: as for outcome 59
Time Frame: 24 months
Population: Of 78 total population, 40 participants were included in the analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 4 patients Mitral Valve Area evaluation was not done or un-evaluable
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 40
cm^2/m^2 | 1.5 (0.5)

61. Secondary Outcome: Mitral Valve Area Index : By Pressure Half-time Formula
Description: as for outcome 59
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 35
cm^2/m^2 | 1.5 (0.5)

62. Secondary Outcome: Mitral Valve Area Index : By Pressure Half-time Formula
Description: as for outcome 59
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 30
cm^2/m^2 | 1.5 (0.5)

63. Secondary Outcome: Mitral Valve Area Index : By Pressure Half-time Formula
Description: as for outcome 59
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
cm^2/m^2 | 1.5 (0.4)

64. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 30 days
Population: Of 78 total population, 69 participants were included in the analysis population because of 6 deaths within 30 days and in 3 participants Mitral Valve Gradient was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 69
mmHg | 3.9 (2.6)

65. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 12 months
Population: Of 78 total population, 53 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 3 patients Mitral Valve Gradient evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
mmHg | 3.6 (2.9)

66. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 24 months
Population: Of 78 total population, 40 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 4 patients Mitral Valve Gradient evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 40
mmHg | 3.2 (1.9)

67. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 36 months
Population: Of 78 total population, 36 participants were included in analysis population because of 31 deaths within 2 years, 7 withdrawals, 1 missed visit and in 3 patients Mitral Valve Gradient evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 36
mmHg | 3.8 (2.7)

68. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 48 months
Population: Of 78 total population, 31 participants were included in analysis population because of 31 deaths within 3 years, 7 withdrawals, 1 missed visit and in 8 patients Mitral Valve Gradient evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
mmHg | 3.6 (1.8)

69. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
mmHg | 3.8 (2)

70. Secondary Outcome: Mitral Valve Index
Description: Mitral valve area as measured by core lab echocardiography and indexed to body surface area [MVA Index = MVA (cm^2)/BSA (m^2)]
Time Frame: 30 days
Population: Of 78 total population, 50 participants were included in the analysis population because of 6 deaths within 30 days and in 22 participants Mitral valve index was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 50
cm^2/m^2 | 1.7 (0.5)

71. Secondary Outcome: Mitral Valve Index
Description: as for outcome 70
Time Frame: 12 months
Population: Of 78 total population, 45 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 11 patients Mitral valve index evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 45
cm^2/m^2 | 1.6 (0.5)

72. Secondary Outcome: Number of Participants With New Coumadin Use
Description: New onset use of Coumadin or warfarin to treat a potential thrombus on a defibrillator lead.
Time Frame: 30 days
Population: 49 patients not on coumadin at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 49
Participants | 9

73. Secondary Outcome: Number of Participants With New Coumadin Use
Description: New onset use of Coumadin or warfarin to treat a potential thrombus on a defibrillator lead.
Time Frame: 6 months
Population: 49 patients not on coumadin at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 49
Participants | 11

74. Secondary Outcome: Number of Participants With New Coumadin Use
Description: New onset use of Coumadin or warfarin to treat a potential thrombus on a defibrillator lead.
Time Frame: 12 months
Population: 49 patients not on coumadin at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 49
Participants | 12

75. Secondary Outcome: Number of Participants Discharged to a Nursing Home or Skilled Nursing Facility or Hospital
Description: Discharge to a nursing home or skilled nursing facility following discharge from the hospital after definitive treatment.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 6

76. Secondary Outcome: Post-procedure Length of Hospital Stay
Description: Defined as the number of days from the end of the procedure until the patient is discharged from the hospital. This does not include time in a nursing or skilled care facility.
Time Frame: Length of Hospital Stay, assessed at 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
days | 3.9 (6.4)

77. Secondary Outcome: Post-procedure Intensive Care Unit (ICU)/ Critical Care Unit (CCU) Time
Description: Number of hours patients are in an intensive care unit or step down unit before discharge or moving to a standard care unit.
Time Frame: Length of ICU/CCU stay, assessed at 30 Days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
hours | 52.3 (80.6)

78. Secondary Outcome: Number of Participants With Successful Clip Implant
Description: Rate of successful delivery and deployment of Clip implants with echocardiographic evidence of leaflet approximation and retrieval of the investigational delivery catheter.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 74

79. Secondary Outcome: Number of Participants With High Risk Procedural Success
Description: Successful implantation of the Clip (s) with resulting MR severity of 2+ of less at discharge or a 1 grade MR reduction at discharge accompanied by a 1 level reduction in NYHA.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 60

80. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity: Site-assessed mitral regurgitation severity using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 1+ to 2+ is mild-to-moderate, 2+ to 3+ is moderate to moderate-to-Severe, 3+ is moderate-to-severe, 3+ to 4+ is moderate-to-severe to severe, 4+ is severe.
Time Frame: Discharge or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 76
Participants
  0 : None | 0
  1+: Mild | 30
  2+: Moderate | 26
  3+: Moderate to Severe | 14
  4+: Severe | 6

81. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 80
Time Frame: 12 months
Population: Of 78 total population, 54 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and MR Severity not done or un-evaluable in 2 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
Participants
  0+: None | 0
  1+: Mild | 17
  2+: Moderate | 25
  3+: Moderate to Severe | 9
  4+: Severe | 3

82. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 80
Time Frame: 24 months
Population: Of 78 total population, 42 participants were included in the analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and MR severity not assessed in 2 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 42
Participants
  0+: None | 0
  1+: Mild | 14
  2+: Moderate | 23
  3+: Moderate to Severe | 5
  4+: Severe | 0

83. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 80
Time Frame: 36 months
Population: Of 78 total population, 37 participants were included in the analysis population because of 31 deaths within 3 years, 7 withdrawals, 1 missed visit and MR Severity was not done or un-evaluable in 2 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 37
Participants
  0+: None | 0
  1+: Mild | 16
  2+: Moderate | 16
  3+: Moderate to Severe | 5
  4+: Severe | 0

84. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 80
Time Frame: 48 months
Population: Of 78 total population, 31 participants were included in the analysis population because of 33 deaths within 3 years, 8 withdrawals, 3 missed visit and MR severity was not done or un-evaluable in 3 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
Participants
  0+: None | 0
  1+: Mild | 18
  2+: Moderate | 9
  3+: Moderate to Severe | 3
  4+: Severe | 1

85. Secondary Outcome: Number of Participants With MR Severity
Description: as for outcome 80
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
Participants
  0+: None | 0
  1+: Mild | 12
  2+: Moderate | 6
  3+: Moderate to Severe | 6
  4+: Severe | 0

86. Secondary Outcome: Number of Participants With Treatment Durability
Description: Defined as the proportion of Acute Procedural Success patients with MR severity grade of 2+ or less that have not required surgery for valve dysfunction.
Time Frame: 12 months
Population: Of 78 total population, 56 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals and 1 missed visit.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 56
Participants | 39

87. Secondary Outcome: Number of Participants With Treatment Durability
Description: as for outcome 86
Time Frame: 24 months
Population: At 24 months, of the 56 patients who achieved acute procedural success, the status of 3 patients is unknown. Among the remaining 53 patients, 30 patients (56.6%) were alive and free from MR > 2+ at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
Participants | 30

88. Secondary Outcome: Number of Participants With Clinical Durability
Description: Proportion of patients who have an acute reduction in MR severity of at least one grade (as measured by the discharge echocardiogram) that have not required surgery for valve dysfunction and meet either of the following: 1) MR severity grade of 2+ or less or 2) a one grade reduction in MR severity compared to baseline accompanied by at least a one level reduction in NYHA.
Time Frame: 12 months
Population: There were 62 patients with an acute reduction in MR severity of at least one grade, and of these, 43 patients met the criterion for clinical durability. The clinical durability rate is therefore 43/62, or 69.4%.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 62
Participants | 43

89. Secondary Outcome: Number of Participants With Clinical Durability
Description: as for outcome 88
Time Frame: 24 months
Population: Through 24 months, the clinical durability status of 3 patients is unknown and there were 35 patients with an acute reduction in MR severity from baseline of at least one grade (the one patient who underwent surgery between 12 months and 24 months is not included in the 35 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 59
Participants | 35

90. Secondary Outcome: Number of Participants With Composite Functional and Structural Measures - Clinical Measures of Benefit-New York Heart Association (NYHA) Class
Description: as for outcome 4
Time Frame: 24 months
Population: Of 78 total population, 43 participants were included in the analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and 1 patient without NYHA Class assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 43
Participants
  NYHA Functional Class I | 13
  NYHA Functional Class II | 24
  NYHA Functional Class III | 5
  NYHA Functional Class IV | 1

91. Secondary Outcome: Number of Participants With Composite Functional and Structural Measures - Clinical Measures of Benefit-New York Heart Association (NYHA) Class
Description: as for outcome 4
Time Frame: 36 months
Population: Of 78 total population, 37 participants were included in analysis population because of 31 deaths within 3 years, 7 withdrawals, 1 missed visit and 2 patients without NYHA Class assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 37
Participants
  NYHA Functional Class I | 10
  NYHA Functional Class II | 20
  NYHA Functional Class III | 7
  NYHA Functional Class IV | 0

92. Secondary Outcome: Number of Participants With Composite Functional and Structural Measures - Clinical Measures of Benefit-New York Heart Association (NYHA) Class
Description: as for outcome 4
Time Frame: 48 months
Population: Of 78 total population, 31 participants were included in the analysis population because of 33 deaths within 3 years, 8 withdrawals, 3 missed visit and NYHA was not assessed in 3 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
Participants
  NYHA Functional Class I | 8
  NYHA Functional Class II | 20
  NYHA Functional Class III | 3
  NYHA Functional Class IV | 0

93. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Class
Description: as for outcome 4
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
Participants
  NYHA Functional Class I | 6
  NYHA Functional Class II | 14
  NYHA Functional Class III | 4
  NYHA Functional Class IV | 0

94. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV).
Description: as for outcome 6
Time Frame: 24 months
Population: Of 78 total population, 39 participants were included in the analysis population because of 26 deaths within 2 year, 7 withdrawals, 1 missed visit and LVEDV was not done or un-evaluable in 5 patients.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
mL | 136.3 (37.8)

95. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV).
Description: as for outcome 6
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 36
mL | 135.7 (40.3)

96. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV).
Description: as for outcome 6
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 29
mL | 139.5 (46.6)

97. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV).
Description: as for outcome 6
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
mL | 133.5 (48.9)

98. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV).
Description: as for outcome 7
Time Frame: 24 months
Population: Of 78 total population, 39 participants were included in the analysis population because of 26 deaths within 2 year, 7 withdrawals, 1 missed visit and LVESV was not done or un-evaluable in 5 patients.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
mL | 71.3 (33.4)

99. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV).
Description: as for outcome 7
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 36
mL | 66.4 (33.1)

100. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV).
Description: as for outcome 7
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 28
mL | 73.3 (36.9)

101. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV).
Description: as for outcome 7
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
mL | 67.2 (38)

102. Secondary Outcome: Left Ventricular Measurement: Left Ventricular Internal Dimension Diastole (LVIDd), Left Ventricular Internal Dimension Systole (LVIDs)
Description: as for outcome 8
Time Frame: 24 months
Population: Of 78 total population, 42 participants were included in the analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and LVIDd/LVIDs not done or un-evaluable in 2 patients.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 42
cm
  LV Internal Diameter, Diastole (LVIDd) | 5.3 (0.8)
  LV Internal Diameter, Systole (LVIDs) | 4.0 (1.0)

103. Secondary Outcome: Left Ventricular Measurement: Left Ventricular Internal Dimension Diastole (LVIDd), Left Ventricular Internal Dimension Systole (LVIDs)
Description: as for outcome 8
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 37
cm
  LV Internal Diameter, Diastole (LVIDd) | 5.4 (0.8)
  LV Internal Diameter, Systole (LVIDs) | 4.1 (1.1)

104. Secondary Outcome: Left Ventricular Measurement: Left Ventricular Internal Dimension Diastole (LVIDd), Left Ventricular Internal Dimension Systole (LVIDs)
Description: as for outcome 8
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
cm
  LV Internal Diameter, Diastole (LVIDd) | 5.5 (0.7)
  LV Internal Diameter, Systole (LVIDs) | 4.0 (1.0)

105. Secondary Outcome: Left Ventricular Measurement: Left Ventricular Internal Dimension Diastole (LVIDd), Left Ventricular Internal Dimension Systole (LVIDs)
Description: as for outcome 8
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
cm
  LV Internal Diameter, Diastole (LVIDd) | 5.5 (0.8)
  LV Internal Diameter, Systole (LVIDs) | 4.2 (1.0)

106. Secondary Outcome: Number of Days Re-hospitalized for CHF
Description: Defined as the number of days hospitalized for CHF in the 12-months prior to the Clip implant procedure date compared to the number of days re-hospitalized for CHF in the 12-months after Clip implant.
Time Frame: 12 months
Population: 12/75 hospitalized for CHF post-discharge, representing 22 separate hospitalization events with mean of 6.6+/-3.7 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 12
days | 6.6 (3.7)

107. Secondary Outcome: Number of Hospital Re-Admissions for Congestive Heart Failure (CHF)
Description: Defined as the number of hospital admissions (i.e. events) for which the primary diagnosis for hospitalization is congestive heart failure, in the 12-months post-discharge following the MitraClip procedure.
Time Frame: 12 months
Population: Of 78 patients, 3 patients who died prior to discharge were not included.
Measure: Number; unit: Events
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
Events | 22

108. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as measured by the core echocardiographic laboratory at follow-up.
Time Frame: 30 days
Population: Of 78 total population, 58 participants were included in the analysis population because of 6 deaths within 30 days and 14 missing data (not done or not evaluable).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 58
mL | 25.2 (14.4)

109. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as measured by the core echocardiographic laboratory at follow-up.
Time Frame: 12 months
Population: Of 78 total population, 44 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 6 patients Regurgitant volume evaluation was not done or not evaluable.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 44
mL | 20.4 (15.4)

110. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as measured by the core echocardiographic laboratory at follow-up.
Time Frame: 24 months
Population: Of 78 total population, 26 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and 18 patients were without Regurgitant Volume assessment.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 26
mL | 19.9 (10.7)

111. Secondary Outcome: Regurgitant Fraction (RF)
Description: RF is defined as the percentage of the left ventricular (LV) stroke volume that regurgitates into the left atrium.
Time Frame: 30 days
Population: Of 78 total population, 58 participants were analysed as 6 participants died within 30 days and 14 missing data (not done or not evaluable).
Measure: Mean (Standard Deviation); unit: percentage of LV stroke volume
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 58
percentage of LV stroke volume | 32.1 (15.2)

112. Secondary Outcome: Regurgitant Fraction
Description: RF is defined as the percentage of the left ventricular (LV) stroke volume that regurgitates into the left atrium.
Time Frame: 12 months
Population: Of 78 total population, 44 participants were included in the analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 6 patients Regurgitant fraction evaluation was not done or not evaluable.
Measure: Mean (Standard Deviation); unit: percentage of LV stroke volume
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 44
percentage of LV stroke volume | 26.3 (16.5)

113. Secondary Outcome: Regurgitant Fraction
Description: RF is defined as the percentage of the left ventricular (LV) stroke volume that regurgitates into the left atrium.
Time Frame: 24 months
Population: Of 78 total population, 26 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and 18 patients were without Regurgitant fraction assessment.
Measure: Mean (Standard Deviation); unit: percentage of LV stroke volume
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 26
percentage of LV stroke volume | 27.4 (13.0)

114. Secondary Outcome: Cardiac Output (CO)
Description: CO is defined as the volume of blood pumped by the left ventricle per unit time (L/min).
Time Frame: 30 Days
Population: Of 78 total population, 66 participants were included in analysis population because of 6 deaths within 30 days and in 6 patients Cardiac Output was not assessed or or un-evaluable.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 66
l/min | 3.8 (1.2)

115. Secondary Outcome: Cardiac Output
Description: CO is defined as the volume of blood pumped by the left ventricle per unit time (L/min)
Time Frame: 12 months
Population: Of 78 total population, 53 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 3 patients Cardiac output evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
l/min | 3.8 (1.0)

116. Secondary Outcome: Cardiac Output
Description: CO is defined as the volume of blood pumped by the left ventricle per unit time (L/min)
Time Frame: 24 months
Population: Of 78 total population, 40 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 4 patients Cardiac output evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 40
l/min | 3.5 (0.9)

117. Secondary Outcome: Cardiac Index
Description: Cardiac index (cardiac output divided by body surface area) as measured by core lab echocardiography.
Time Frame: 30 Days
Population: Of 78 total population, 66 participants were included in the analysis population because of 6 deaths within 30 days and in 6 participants cardiac Index was un-evaluable or not done.
Measure: Mean (Standard Deviation); unit: l/min/m2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 66
l/min/m2 | 2 (0.6)

118. Secondary Outcome: Cardiac Index
Description: Cardiac index (cardiac output divided by body surface area) as measured by core lab echocardiography.
Time Frame: 12 months
Population: Of 78 total population, 53 participants were included in analysis population because of 18 deaths within 1 year, 3 withdrawals, 1 missed visit and in 3 patients Cardiac Index evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: l/min/m2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 53
l/min/m2 | 2 (0.5)

119. Secondary Outcome: Cardiac Index
Description: Cardiac index (cardiac output divided by body surface area) as measured by core lab echocardiography.
Time Frame: 24 months
Population: Of 78 total population, 40 participants were included in analysis population because of 26 deaths within 2 years, 7 withdrawals, 1 missed visit and in 4 patients cardiac index evaluation was not done or un-evaluable.
Measure: Mean (Standard Deviation); unit: l/min/m2
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 40
l/min/m2 | 1.8 (0.4)

120. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: Discharge or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
percentage of ejection fraction | 52.3 (12.4)

121. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 54
percentage of ejection fraction | 50.2 (13.1)

122. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
percentage of ejection fraction | 49.5 (12)

123. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 36
percentage of ejection fraction | 52.5 (12.5)

124. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 28
percentage of ejection fraction | 49.9 (12.6)

125. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as determined by the core echocardiography laboratory.
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 24
percentage of ejection fraction | 51.5 (13.6)

126. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: Percentage of patients who did not undergo surgical mitral valve repair or replacement after the index MitraClip procedure
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
percentage of participants | 100

127. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: as for outcome 126
Time Frame: 12 months
Population: Analysis population includes 58 participants, which represents the number of patients at risk as per Kaplan-Meier freedom from Mitral valve (MV)surgery analysis at 12 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 58
percentage of participants | 100

128. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: as for outcome 126
Time Frame: 24 months
Population: Analysis population includes 45 participants, which represents the number of patients at risk as per Kaplan-Meier analysis at 24 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 45
percentage of participants | 98.1

129. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: as for outcome 126
Time Frame: 36 months
Population: Analysis population includes 39 participants, which represents the number of patients at risk as per Kaplan-Meier analysis at 36 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
percentage of participants | 98.1

130. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: as for outcome 126
Time Frame: 48 months
Population: Analysis population includes 35 participants, which represents the number of patients at risk as per Kaplan-Meier analysis at 48 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 35
percentage of participants | 95.5

131. Secondary Outcome: Percentage of Participants With Freedom From Mitral Valve Surgery
Description: as for outcome 126
Time Frame: 60 months
Population: Analysis population includes 14 participants, which represents the number of patients at risk as per Kaplan-Meier analysis at 60 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 14
percentage of participants | 95.5

132. Secondary Outcome: Number of Participants With Mitral Valve Repair Success
Description: Mitral Valve Repair Success defined as freedom from mitral valve replacement surgery for valve dysfunction, death, re-operation and MR > 2+ at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 44

133. Secondary Outcome: Number of Participants With Mitral Valve Repair Success
Description: Freedom from mitral valve replacement surgery for Valve Dysfunction, death, re-operation, and MR > 2+.
Time Frame: 24 months
Population: Three Acute Procedural Success (APS) patients withdrew at or before 12 months, and had MR ≤ 2+ at all visits prior to withdrawal. Since there is no data on these patients post-12 months, these patients are not included in the endpoint of freedom from mitral valve replacement surgery for Valve Dysfunction, death and MR > 2+ at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
Participants | 37

134. Secondary Outcome: Composite Functional and Structural Measures - Percentage of Participants With Freedom From Death
Description: as for outcome 1
Time Frame: 24 months
Population: Analysis population includes 46 participants, which represents the number of patients at risk as per Kaplan-Meier freedom from mortality analysis at 24 months.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 46
percentage of participants | 64.6

135. Secondary Outcome: Percentage of Participants With Composite Functional and Structural Measures - Freedom From Death and MR >2+
Description: Kaplan-Meier estimated proportion of patients who are alive and have a mitral regurgitation severity grade of 2+ or less.
Time Frame: 24 months
Population: Primary Analysis at 24 months included only 75 patients. Three patients were excluded due to withdrawal at or before 12 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
percentage of participants
  Primary Analysis: number analyzed (Participants) | 75
  Primary Analysis | 49.3 [37.6 to 61.1]
  Worstcase Analysis | 46.2 [34.8 to 57.8]

136. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment
Description: Device embolization is defined as bilateral Clip detachment resulting in Clip embolization. Reasons for Clip embolization include leaflet tearing, Clip unlocking, Clip fracture or inadequate Clip placement (i.e., malposition). Not included are any fractures or other failures of the Clip that do not result in Clip detachment from both leaflets.
  A single leaflet device attachment (SLDA) is defined as attachment of one mitral valve leaflet to the MitraClip device.
Time Frame: 0 to 12 months
Population: Three patients were excluded from the analysis as they did not receive a Device.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 75
Participants
  Device Embolization | 0
  Single Leaflet Device Attachment | 1

137. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment
Description: as for outcome 136
Time Frame: 24 months
Population: Patients implanted with a MitraClip device, alive were evaluated at 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 46
Participants
  Device Embolization | 0
  Single Leaflet Device Attachment | 0

138. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment
Description: as for outcome 136
Time Frame: 48 months
Population: Patients implanted with a MitraClip device and alive were evaluated at 48 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 31
Participants
  Device Embolization | 0
  Single Leaflet Device Attachment | 0

139. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment
Description: as for outcome 136
Time Frame: 36 months
Population: Patients implanted with a MitraClip device, alive were evaluated at 36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
Participants
  Device Embolization | 0
  Single Leaflet Device Attachment | 0

140. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment
Description: as for outcome 136
Time Frame: 60 months
Population: Patients implanted with a MitraClip device and alive were evaluated at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 30
Participants
  Device Embolization | 0
  Single Leaflet Device Attachment | 0

141. Secondary Outcome: Number of Participants With Mitral Valve Surgery Post-MitraClip Procedure
Description: Number of patients who underwent surgical mitral valve repair or replacement after the index MitraClip procedure.
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 30
Participants | 2

142. Secondary Outcome: Number of Participants With Second MitraClip Device Implanted
Description: It is a summary of re-interventions to place an additional MitraClip Device.
Time Frame: 0 to 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 30
Participants | 2

143. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality and Mitral Valve Surgery
Description: Kaplan-Meier estimate of the percentage of patients who are alive and did not undergo surgical mitral valve repair or replacement after the index MitraClip procedure
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 58
percentage of participants | 75.6

144. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality and Mitral Valve Surgery
Description: as for outcome 143
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 45
percentage of participants | 63.2

145. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality and Mitral Valve Surgery
Description: as for outcome 143
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 39
percentage of participants | 57.4

146. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality and Mitral Valve Surgery
Description: as for outcome 143
Time Frame: 48 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 35
percentage of participants | 51.5

147. Secondary Outcome: Percentage of Participants With Freedom From All-Cause Mortality and Mitral Valve Surgery
Description: as for outcome 143
Time Frame: 60 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 14
percentage of participants | 41.2

148. Secondary Outcome: Number of Participants With Mitral Valve Replacement
Description: Defined as how often patients receiving surgery required replacement of the mitral valve.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

149. Secondary Outcome: Number of Participants With Mitral Valve Replacement
Description: Defined as how often patients receiving surgery required replacement of the mitral valve.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 1

150. Secondary Outcome: Number of Participants With Mitral Valve Replacement
Description: Defined as how often patients receiving surgery required replacement of the mitral valve.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

151. Secondary Outcome: Number of Participants With Mitral Valve Replacement
Description: Defined as how often patients receiving surgery required replacement of the mitral valve.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Registry Arm
Number analyzed (Participants) | 78
Participants | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | High Risk Registry Arm
All-Cause Mortality (participants affected / at risk) | 25/78
Serious Adverse Events (participants affected / at risk) | 69/78
Other Adverse Events (participants affected / at risk) | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Registry Arm (N=78)
Anemia (Blood and lymphatic system disorders) | 9
Coagulopathy (Blood and lymphatic system disorders) | 2
Hematologic - Other (Blood and lymphatic system disorders) | 2
Infection/Bacteremia/Septicemia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial arrhythmia (Cardiac disorders) | 9
Atrial septal defect (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 3
Cardiac disorders: Other (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Chest pain/Angina (Cardiac disorders) | 9
Congestive heart failure (Cardiac disorders) | 21
Coronary artery disease (Cardiac disorders) | 2
Endocarditis (Cardiac disorders) | 2
Heart block (Cardiac disorders) | 3
Lead displacement (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 7
Myocardial ischemia (Cardiac disorders) | 1
Other rhythm disorder (Cardiac disorders) | 7
Palpitations (Cardiac disorders) | 1
Residual/Recurrent MR (Cardiac disorders) | 1
Supraventricular arrhythmia (Cardiac disorders) | 1
Syncope/Dizziness (Cardiac disorders) | 2
Tamponade (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Bleed (Gastrointestinal disorders) | 9
Gastrointestinal disorders: Other (Gastrointestinal disorders) | 9
Infection (Gastrointestinal disorders) | 1
Death (General disorders) | 25
General disorders: Other (General disorders) | 11
Generalized weakness/Fatigue (General disorders) | 2
Infection (General disorders) | 7
Metabolic/Endocrine disorders (General disorders) | 7
Connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8
Intracerebral hemorrhage (Nervous system disorders) | 5
Nervous system disorders: Other (Nervous system disorders) | 6
Neurologic - Stroke (Nervous system disorders) | 1
Transient ischemic attack (TIA) (Nervous system disorders) | 6
Renal Infection (Renal and urinary disorders) | 9
Renal and urinary disorders: Other (Renal and urinary disorders) | 2
Renal insufficiency/Failure (Renal and urinary disorders) | 20
Bronchial/lung disorders (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 11
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11
Arteriovenous (AV) fistula (Vascular disorders) | 2
Bleeding complication (Vascular disorders) | 5
Deep vein thrombosis (DVT) (Vascular disorders) | 1
Embolization (Vascular disorders) | 1
Hemodynamic instability (Vascular disorders) | 9
Pseudoaneurysm (Vascular disorders) | 2
Shock (Vascular disorders) | 1
Vascular Injury (Vascular disorders) | 1
Vascular disorders: Other (Vascular disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Registry Arm (N=78)
Anemia (Blood and lymphatic system disorders) | 26
Hemolysis (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Atrial arrhythmia (Cardiac disorders) | 10
Atrial septal defect (Cardiac disorders) | 4
Bradyarrhythmia (Cardiac disorders) | 4
Cardiac disorders: other (Cardiac disorders) | 4
Chest pain/Angina (Cardiac disorders) | 22
Congestive heart failure (Cardiac disorders) | 19
Myocardial ischemia (Cardiac disorders) | 9
Other rhythm disorder (Cardiac disorders) | 8
Peripheral edema (Cardiac disorders) | 20
Residual/recurrent magnetic resonance (MR) (Cardiac disorders) | 15
Syncope/Dizziness (Cardiac disorders) | 19
Ventricular arrhythmia (Cardiac disorders) | 6
cardiomyopathy (Cardiac disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 4
Bleed (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 8
Gastrointestinal disorders: Other (Gastrointestinal disorders) | 30
Infection (Gastrointestinal disorders) | 8
Fever (General disorders) | 6
General disorders: Other (General disorders) | 38
Generalized weakness/Fatigue (General disorders) | 24
Incisional site pain (General disorders) | 13
Infection (General disorders) | 6
Mental disorders (General disorders) | 14
Metabolic/Endocrine disorders (General disorders) | 26
Skin/Mucosal/Subcutaneous tissue disorders (General disorders) | 10
Connective tissue disorders (Musculoskeletal and connective tissue disorders) | 37
Nervous system disorders: Other (Nervous system disorders) | 18
Transient ischemic attack (TIA) (Nervous system disorders) | 4
Renal Infection (Renal and urinary disorders) | 10
Renal and urinary disorders: Other (Renal and urinary disorders) | 12
Renal insufficiency/Failure (Renal and urinary disorders) | 15
Bronchial/Lung disorders (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory, thoracic and mediastinal disorders: Other (Respiratory, thoracic and mediastinal disorders) | 30
Bleeding complication (Vascular disorders) | 34
Blood pressure complication (Vascular disorders) | 4
Bruise/Contusion/Ecchymosis (Vascular disorders) | 18
Hematoma (Vascular disorders) | 19
Hemodynamic instability (Vascular disorders) | 21
Vascular disorders: Other (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days